CLINICAL TRIAL: NCT01077895
Title: The Influence of Fluid Removal Using Continuous Venovenous Hemofiltration (CVVH) on Intra-abdominal Pressure and Kidney Function in Critically Ill Adults With Intra-abdominal Hypertension and Acute Kidney Injury
Brief Title: The Influence of Fluid Removal Using Continuous Venovenous Hemofiltration (CVVH) on Intra-abdominal Pressure and Kidney Function
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Stuivenberg Hospital Antwerp (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2009/721
Record Dates: First submitted 2010-02-25; First posted 2010-03-01 (Estimated); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Critically Ill; Intra-Abdominal Hypertension; Abdominal Compartment Syndrome; Acute Kidney Injury
Keywords: Critically ill patients with positive fluid balance, IAH and AKI requiring RRT
MeSH Terms: conditions — Critical Illness; Intra-Abdominal Hypertension; Acute Kidney Injury | interventions — Ultrafiltration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- CVVH with fluid removal (Experimental)
  Interventions: Procedure: CVVH; Procedure: ultrafiltration
- CVVH without fluid removal (Active Comparator)
  Interventions: Procedure: CVVH; Procedure: ultrafiltration control group

INTERVENTIONS:
Procedure: CVVH — CVVH is started using following parameters:
  * Blood flow is started at 150 mL/min
  * Anticoagulation: none, heparin or low molecular weight heparin according to local protocols in study centers.
  * In both groups: dialysis dose of 25 mL/kg body weight administered using both pre- and postdilution
  * Substitution fluid temperature is started at 37°C and adjusted in function of patient body temperature (which is maintained at 35-37°C)
Procedure: ultrafiltration — ultra filtration is started at 100 mL/h and increased according to following protocol
  * Ultrafiltration is increased by 100 mL/h after 2h and subsequently by 100mL/h (until a maximum of 500mL/h) every 4h unless:
  * Vasopressor or inotrope medication dose is increased by > 25% (provided mean arterial pressure remains constant at 65 mmHg or another target value specified by treating physician according to standard of care)
  * When above condition is not met UF should be kept constant and a passive leg raising test or stroke volume variation measurement should be performed. If SVV > 10% or PLR is positive 100mL of albumin 20% solution or 250 mL of Hydroxyethyl Starch 130/0.4 solution is administered according to treating physician at a maximum of 4 times per 24h
  * If there is no improvement after 2 colloid administration rounds, UF should be stopped for 4h and restarted at half the rate it was set at when discontinued.
  Arms: CVVH with fluid removal
Procedure: ultrafiltration control group — ultrafiltration is set at 100 mL/h (and fluid administration is titrated to approach 100 mL /h)
  Arms: CVVH without fluid removal

SUMMARY:
Intra- abdominal hypertension (IAH) and abdominal compartment syndrome (ACS) are a cause of organ dysfunction in critically ill patients. IAH develops due to abdominal lesions (primary IAH) or extra-abdominal processes (secondary IAH). Secondary IAH arises due to decreased abdominal wall compliance and gut edema caused by capillary leak and excessive fluid resuscitation. Decreasing intra-abdominal pressure (IAP) using decompressieve laparotomy has been shown to improve organ dysfunction. However, laparotomy is generally avoided in patients with secondary IAH due to the risk of abdominal complications.

Acute kidney injury (AKI) is one of the first and most pronounced organ failures associated with IAH and many patients with AKI in the ICU require renal replacement therapy (RRT). Fluid removal using continuous RRT (CRRT) has been demonstrated to decrease IAP in small series and selected patients.

The aim of this study is to evaluate whether fluid removal using CVVH in patients with IAH, fluid overload and AKI is feasible and whether it has a beneficial effect on organ dysfunction (compared to CVVH without net fluid removal).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18y old) of either gender
* Admitted to the ICU
* Sedated and mechanically ventilated (and expected to remain so for at least 48h)
* Informed consent given
* admitted to the ICU for <7 days or during the first 7 days of a new shock episode
* AKI requiring RRT according to treating physician
* IAP >12mmHg being attributed to fluid overload by treating physician

Exclusion Criteria:

* Included in the same study before
* Vasopressor and/or inotrope dose needed above noradrenaline 1µg/kg/min and dobutamine 10µg/kg/min
* PaO2/FiO2 ratio <100

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Change in IAP in patients receiving fluid removal during CVVH vs patients receiving CVVH without net fluid removal after 24 and 48h of CVVH treatment | 24 and 48 hours

SECONDARY OUTCOMES:
Difference between CVVH with fluid removal and CVVH without fluid removal | after 24 hours and/or 7 days
  Difference in terms of
  * Need for vasopressor medication and hemodynamic parameters during the first seven days
  * PaO2/FiO2 (worst value over 24h daily first 7 days)
  * Volume of albumin solution or synthetic colloids administered during CVVH per 24h
  * SOFA score daily first seven days
  * Need for decompressive laparotomy or other means to decrease IAP
  * Acid-base status
  * Complications relating to ischemia
Difference between both groups in terms of daily fluid balance | during 7 days
The relationship between cumulative fluid balance at the start of each day of CVVH and the fluid balance achieved after 24h of CVVH with fluid removal | 24 hours
Difference between both groups regarding recovery of renal function, need for RRT at discharge from the ICU and from the hospital | discharge from ICU and hospital
Difference between both groups regarding mortality (28d, ICU and hospital) and ICU and hospital length of stay | 28 days and length of stay in ICU and hospital

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hoste, MD, Phd, Principal Investigator — University Hospital Ghent, Belgium
Locations (2):
- Belgium (2):
  - ZNA Stuivenberg Hospital, Antwerp
  - University Hospital Ghent, Ghent

REFERENCES:
- See also: website of the University Hospital Ghent — http://www.uzgent.be